CLINICAL TRIAL: NCT03935542
Title: Anatomical Attributes of Clinically Relevant Diagonal Branches in Patients With Left Anterior Descending Coronary Artery Bifurcation Lesions
Brief Title: Assessment of Diagonal Branch Territory
Status: Completed | Type: Observational
Sponsor: Bon-Kwon Koo (Other)
Collaborators: Seoul National University Hospital (Other); Naju National Hospital (Other); Chonnam National University Hospital (Other); Samsung Medical Center (Other); Ewha Womans University (Other); Ajou University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Other Study IDs: SB-FMM-prediction
Record Dates: First submitted 2019-04-26; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Stable Angina; Unstable Angina
Keywords: Bifurcation; Side branch; Ischemia; Myocardium; Revascularization
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- MPI arm: For the MPI arm, patients with severe jailed diagonal branch disease with available MPI in 3 months were selected from the Seoul National University Hospital Cardiac Catheterization and MPI database.
- CCTA arm: For the CCTA arm, patients from a previous multicenter prospective CCTA registry were retrospectively reviewed for a post-hoc analysis.

SUMMARY:
This study was performed to investigate the anatomical attributes that determine myocardial territory of diagonal branches and to develop a prediction model for clinically relevant branches using myocardial perfusion imaging (MPI) and coronary CT angiography (CCTA).

DETAILED DESCRIPTION:
Bifurcation lesion is one of the most challenging lesion subsets in the field of percutaneous coronary intervention (PCI). Despite the recent advances in PCI techniques and stent technology, most randomized studies failed to prove the superiority of systematic 2 stenting strategy compared with provisional side branch intervention strategy.

A certain amount of ischemic burden is required to achieve the benefit of revascularization over medical treatment. Compared with major epicardial vessels, side branches are smaller, more variable in anatomy, supplying less myocardium and less clinically relevant. Therefore, it is important to assess the myocardial mass at risk of side branches to determine the appropriate treatment strategy for bifurcation lesions. However, how to define the clinically relevant side branches which can be associated with the benefit of revascularization in a cardiac catheterization laboratory is not well-known.

The investigators performed this study to investigate the anatomical attributes that determine ischemic burden and myocardial territory of diagonal branches and to develop a prediction model for a clinically relevant diagonal branch using myocardial perfusion imaging (MPI) and coronary CT angiography (CCTA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe jailed diagonal branch disease with available MPI in 3 months (MPI arm)
* Patients who had available FMM value of diagonal branches from a previous multicenter prospective CCTA registry (CCTA arm)

Exclusion Criteria:

* Patients with >50% stenosis at left anterior descending coronary artery (LAD) or left circumflex artery (LCx), regional wall motion abnormality at LAD territory (MPI arm)
* Patients with diffuse diagonal branch disease (CCTA arm)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with angina pectoris
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Angiographic attributes for diagonal branches | through study completion, an average of 1year
  Angiographic attributes for diagonal branches were visually defined as follows :
  1. Size was a binary attribute of vessel diameter ≥ 2.5mm or < 2.5mm.
  2. Number was counted as one, two, and 3 or more diagonal branches.
  3. Dominancy in patients with 2 diagonal branches (D1/2 dominancy) was a binary attribute for one of two diagonal branches whose diameter was more than two times larger than its smaller counterpart.
  4. LCx dominancy was defined as a left-dominant system or a presence of obtuse marginal branch originating within proximal 1/3 of LCx and crossing LAD at right anterior oblique caudal view.
Sensitivity of prediction model | through study completion, an average of 1year
  Prediction model using anatomical attributes to define clinical relevance of diagonal branches will be developed.
Specificity of prediction model | through study completion, an average of 1year
  Prediction model using anatomical attributes to define clinical relevance of diagonal branches will be developed.
Negative predictive value of prediction model | through study completion, an average of 1year
  Prediction model using anatomical attributes to define clinical relevance of diagonal branches will be developed.
Positive predictive value of prediction model | through study completion, an average of 1year
  Prediction model using anatomical attributes to define clinical relevance of diagonal branches will be developed.
Area under the curve of prediction model | through study completion, an average of 1year
  Prediction model using anatomical attributes to define clinical relevance of diagonal branches will be developed.
Accuracy of prediction model | through study completion, an average of 1year
  Prediction model using anatomical attributes to define clinical relevance of diagonal branches will be developed.

SECONDARY OUTCOMES:
%Ischemia | through study completion, an average of 1year
  Myocardium of perfusion image was divided into 20 segments, and summed rest score (SRS), summed stress score (SSS), and summed difference score (SDS) were scored in each segment according to a 5-grade system (0-4) for the assessment of perfusion status. (1) SSS and SDS of diagonal segments were converted to percent of myocardial ischemia (%ischemia) of diagonal territory by dividing summed scores by 80 and multiplying by 100.
%FMM | through study completion, an average of 1year
  FMM was calculated using stem-and-crown model as described in the parent study. (2) FMM of each diagonal brach was converted to percent FMM (%FMM) of diagonal branch by dividing each FMM by left ventricular myocardial mass.

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Paeng JC, Lee DS, Cheon GJ, Lee MM, Chung JK, Lee MC. Reproducibility of an automatic quantitation of regional myocardial wall motion and systolic thickening on gated 99mTc-sestamibi myocardial SPECT. J Nucl Med. 2001 May;42(5):695-700. PMID 11337562
- [Background] Kim HY, Lim HS, Doh JH, Nam CW, Shin ES, Koo BK, Yoon MH, Tahk SJ, Kang DK, Song YB, Hahn JY, Choi SH, Gwon HC, Lee SH, Kim EK, Kim SM, Choe Y, Choi JH. Physiological Severity of Coronary Artery Stenosis Depends on the Amount of Myocardial Mass Subtended by the Coronary Artery. JACC Cardiovasc Interv. 2016 Aug 8;9(15):1548-60. doi: 10.1016/j.jcin.2016.04.008. Epub 2016 Jul 13. PMID 27423225
- [Derived] Jeon WK, Park J, Koo BK, Suh M, Yang S, Kim HY, Lee JM, Kim KJ, Choi JH, Lim HS, Paeng JC, Hwang D, Kim HS; Collaborators. Anatomical attributes of clinically relevant diagonal branches in patients with left anterior descending coronary artery bifurcation lesions. EuroIntervention. 2020 Oct 9;16(9):e715-e723. doi: 10.4244/EIJ-D-19-00534. PMID 31719001